CLINICAL TRIAL: NCT00284622
Title: A Randomized Clinical Trial to Compare the Effectiveness of High Tibial Osteotomy With or Without Arthroscopy of the Knee Joint on Quality of Life, Functional Ability and Pain for Patients With Medical Compartment Osteoarthritis of the Knee
Brief Title: HTO With and Without Arthroscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Responsible Party: Robert Giffin, FKSMC
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HTO-1
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Medial Compartment Osteoarthritis of the Knee
Keywords: HTO; Arthroscopy; Osteoarthritis; Alignement; Varus gonarthrosis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Procedure: Arthroscopy — HTO with pre-scope

SUMMARY:
It remains unknown if a concomitant arthroscopic knee debridement would increase the benefits of surgery (quality of life and functional ability) for young active patients with medial compartment OA of the knee and varus alignmen. This additional procedure has a low incidence of morbidity and would potentially allow for treatment of meniscal tears and articular damage, as well as joint lavage to remove debris and inflammatory factors. A trial is needed to determine whether HTO with concomitant knee arthroscopy will result in better overall outcomes for this patient group.The objective is to compare the quality of life, functional status, pain, and swelling of patients who undergo an HTO with or without a concomitant knee joint arthroscopy to address additional joint pathology

DETAILED DESCRIPTION:
Arthroscopy for degenerative conditions of the knee is among the most widely employed orthopaedic procedures, but its effectiveness (like the effectiveness of many surgical operations) has never been proven in prospective trials. The evidence supporting the use of arthroscopy in treatment algorithms for knee OA comes largely from case series and cohort studies. These studies have shown that about 50% of patients report pain relief following the procedure. Predictors of poor outcome following arthroscopy include marked mal-alignment, restricted range of motion, advanced radiographic changes, and prior surgery. Improved outcomes are predicted by preoperative mechanical symptoms caused by loose bodies, meniscal tears, or radiographic evidence of mild articular degeneration.

The proposed study is a randomized clinical trial.

Each patient will undergo a preoperative MRI of their affected knee joint to identify existing pathology (e.g. meniscal tears, loose bodies, chondral flaps). The results of the MRI will not be revealed to physicians, patients or data collectors. This will ensure that we have information on the existing joint pathology within each group and that prognostic variables between groups were sufficiently balanced (i.e. comparable rates of similar pathology per group). The primary outcome measure is self-reported quality of life (WOMAC). Secondary measures include self-reported functional ability (LEFS), swelling, pain and frequency of analgesic use (patient diary), and general health (SF-36). Assessments will take place preoperatively and at 3, 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients with medial compartment osteoarthritis as determined by clinical examination and plain radiographs.
* scheduled for an HTO

Exclusion Criteria:

1. Evidence of other significant knee pathology,
2. Active joint or systemic infection,
3. Major medical illness that would preclude undergoing surgery,
4. Patients who are unwilling or unable to be assessed according to study protocol for one year following surgery
5. Major psychiatric illness, developmental handicap or inability to read and understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
self-reported quality of life (WOMAC). | 2 years

SECONDARY OUTCOMES:
self-reported functional ability (LEFS), | 2 years
swelling | 2 years
pain | 2 yrs
frequency of analgesic use (patient diary), | 3 mths
general health (SF-36). | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: J. Robert Giffin, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada